CLINICAL TRIAL: NCT01592695
Title: Tailored Tobacco Cessation Program for Rural Veterans With Comorbid Depression, Alcoholism or Obesity
Brief Title: Tailored Tobacco Quitline for Rural Veterans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iowa City Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark Vander Weg, Research Specialist, Iowa City Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201203712
Record Dates: First submitted 2012-04-11; First posted 2012-05-07 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Cigarette Smoking
Keywords: Nicotine dependence; Smoking cessation; Telehealth; Alcohol use; Depression; Body weight
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder; Smoking Cessation; Alcohol Drinking; Depression; Body Weight | interventions — Bupropion; Varenicline; Nicotine Chewing Gum; Tobacco Use Cessation Devices; Ethanol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored Intervention Group (Experimental): Participants will receive a combined behavioral and pharmacological intervention. The behavioral component will consist of a six-session cognitive behavioral telephone intervention combined with supplemental treatment modules to address common issues associated with cigarette smoking.
  Interventions: Drug: Nicotine replacement therapy - transdermal nicotine patch; Behavioral: Tailored behavioral intervention; Drug: Nicotine replacement therapy - nicotine gum; Drug: Nicotine replacement therapy - nicotine lozenge; Drug: Bupropion Sustained Release; Drug: Varenicline; Drug: Combination pharmacotherapy - transdermal nicotine patch + nicotine gum; Drug: Combination pharmacotherapy - transdermal nicotine patch + nicotine lozenge; Drug: Combination pharmacotherapy - transdermal nicotine patch + bupropion; Behavioral: Alcohol use risk reduction; Behavioral: Behavioral activation for the treatment of depression; Behavioral: Behavioral management of post-cessation weight gain
- Enhanced Standard of Care Group (Active Comparator): Participants assigned to the enhanced standard of care condition will receive referral to their state tobacco quit line along with pharmacotherapy to assist with smoking cessation.
  Interventions: Drug: Nicotine replacement therapy - transdermal nicotine patch; Behavioral: Tobacco quit line referral; Drug: Nicotine replacement therapy - nicotine gum; Drug: Nicotine replacement therapy - nicotine lozenge; Drug: Bupropion Sustained Release; Drug: Varenicline; Drug: Combination pharmacotherapy - transdermal nicotine patch + nicotine gum; Drug: Combination pharmacotherapy - transdermal nicotine patch + nicotine lozenge; Drug: Combination pharmacotherapy - transdermal nicotine patch + bupropion

INTERVENTIONS:
Drug: Nicotine replacement therapy - transdermal nicotine patch — Medication selection will be determined based on individual participant preferences, medical history, and contraindications.
Behavioral: Tailored behavioral intervention — Participants will receive a standard six session cognitive behavioral intervention for smoking cessation combined with supplemental treatment modules based on individual need and preference.
  Arms: Tailored Intervention Group
Behavioral: Tobacco quit line referral — Participants assigned to this condition will receive a referral to their state tobacco quit line. The specific behavioral treatment that is provided will differ slightly depending upon the services available through the participant's state of residence.
  Arms: Enhanced Standard of Care Group
Drug: Nicotine replacement therapy - nicotine gum — Medication selection will be determined based on individual participant preferences, medical history, and contraindications
Drug: Nicotine replacement therapy - nicotine lozenge — Medication selection will be determined based on individual participant preferences, medical history, and contraindications
Drug: Bupropion Sustained Release — Medication selection will be determined based on individual participant preferences, medical history, and contraindications
  Other Names: Zyban
Drug: Varenicline — Medication selection will be determined based on individual participant preferences, medical history, and contraindications
  Other Names: Chantix
Drug: Combination pharmacotherapy - transdermal nicotine patch + nicotine gum — Medication selection will be determined based on individual participant preferences, medical history, and contraindications
Drug: Combination pharmacotherapy - transdermal nicotine patch + nicotine lozenge — Medication selection will be determined based on individual participant preferences, medical history, and contraindications
Drug: Combination pharmacotherapy - transdermal nicotine patch + bupropion — Medication selection will be determined based on individual participant preferences, medical history, and contraindications
Behavioral: Alcohol use risk reduction — Participants engaging in risky alcohol use may receive this six-session telephone-based behavioral intervention for reducing alcohol use.
  Other Names: Risky alcohol use; Harm reduction
  Arms: Tailored Intervention Group
Behavioral: Behavioral activation for the treatment of depression — Participants with elevated depressive symptoms may receive this six-session telephone-based behavioral activation intervention.
  Other Names: Depression
  Arms: Tailored Intervention Group
Behavioral: Behavioral management of post-cessation weight gain — Participants with concerns about gaining weight after quitting smoking may receive this six-session telephone-based behavioral self-management intervention designed to help attenuate post-cessation weight gain.
  Other Names: Weight management
  Arms: Tailored Intervention Group

SUMMARY:
The proposed work is designed to help increase access to tobacco cessation services among rural veterans and to develop more effective treatment services that better address comorbid issues commonly experienced by rural smokers. The objectives are:

1. Study the feasibility of an individually-tailored telephone intervention for rural smokers.
2. Examine the impact of the intervention on tobacco use outcomes.
3. Evaluate the effect of the intervention on issues commonly experienced by rural smokers including depressive symptoms, alcohol use, and weight gain.

DETAILED DESCRIPTION:
Tobacco use remains the leading preventable cause of morbidity and mortality in our society. Results from epidemiologic studies indicate that tobacco use is especially elevated among those living in rural areas. Although interventions exist that are both effective and cost-effective, few rural smokers utilize them during any given quit attempt. A lack of local treatment resources, the travel distance required to obtain treatment, and a reduced tendency to visit primary care on a regular basis all appear to contribute to the lower levels of treatment for nicotine dependence in rural smokers.

Smokers frequently experience conditions and concerns that adversely impact their ability to quit smoking. Depression and risky alcohol use, both of which are prevalent among smokers, reduce the likelihood of successfully quitting smoking. Concern about gaining weight, a common consequence of quitting smoking, is also frequently cited by smokers as an important barrier to quitting. Therefore, in order to be most effective, tobacco cessation interventions will need to address these important issues. Presently, treatment for nicotine dependence, risky alcohol use, depression, and weight management is typically delivered separately and without optimal integration among providers, an approach which only serves to fragment care and increase the number of required visits, further reduce rural smokers' access to care.

In an effort to address these barriers, the current study will evaluate a telephone intervention for tobacco use that also addresses issues related to risky alcohol use, depressed mood, and postcessation weight gain based on each individual smoker's needs. Results will provide valuable information regarding the potential to more widely implement an individually-tailored telephone intervention for rural smokers.

ELIGIBILITY:
Inclusion Criteria:

* Being a veteran
* 18 + years of age
* Smoke cigarettes on at least a daily basis
* Receive primary care from the Iowa City VAMC or Coralville Clinic
* Live in a non-metropolitan area (based on RUCA codes)
* Be willing to make a quit attempt in the next 30 days
* Be capable of providing informed consent
* Have access to a telephone (land line or cell phone)
* Have a stable residence

Exclusion Criteria:

* Planning to move within the next 12 months
* Presence of a terminal illness
* Pregnancy
* Unstable psychiatric disorder (e.g., acute psychosis)
* Currently pregnant
* Incarcerated
* Institutionalized

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark VanderWeg, PhD, Principal Investigator — VRHRC-CR
Locations (1):
- Iowa City VA Health Care System, Iowa City, Iowa, United States

REFERENCES:
- [Result] Vander Weg MW, Cozad AJ, Howren MB, Cretzmeyer M, Scherubel M, Turvey C, Grant KM, Abrams TE, Katz DA. An individually-tailored smoking cessation intervention for rural Veterans: a pilot randomized trial. BMC Public Health. 2016 Aug 17;16(1):811. doi: 10.1186/s12889-016-3493-z. PMID 27535024
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Groups:
- Tailored Intervention Group: Participants will receive a combined behavioral and pharmacological intervention.
  Pharmacotherapy: Medication selection will be determined based on individual participant preferences, medical history, and contraindications. Options will include nicotine replacement therapy (nicotine patch, nicotine gum, nicotine lozenge), bupropion, or varenicline. Medications will be provided as mono-therapy or in combination.
  Tailored behavioral intervention: Participants will receive a standard six session cognitive behavioral intervention for smoking cessation combined with supplemental treatment modules treatment modules to address common issues associated with cigarette smoking based on individual need and preference. Individual treatment models address alcohol risk reduction, elevated depressive symptoms, and concerns about weight gain.
- Enhanced Standard of Care Group: Participants assigned to the enhanced standard of care condition will receive referral to their state tobacco quit line along with pharmacotherapy to assist with smoking cessation.
  Pharmacotherapy: Medication selection will be determined based on individual participant preferences, medical history, and contraindications. Options will include nicotine replacement therapy (nicotine patch, nicotine gum, nicotine lozenge), bupropion, or varenicline. Medications will be provided as mono-therapy or in combination.
  Tobacco quit line referral: Participants assigned to this condition will receive a referral to their state tobacco quit line. The specific behavioral treatment that is provided will differ slightly depending upon the services available through the participant's state of residence.
Period: Overall Study
Arm/Group | Tailored Intervention Group | Enhanced Standard of Care Group
Started | 31 | 32
Completed | 23 | 28
Not Completed | 8 | 4
Not completed — Lost to Follow-up | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Tailored Intervention Group: Participants will receive a combined behavioral and pharmacological intervention.
  Pharmacotherapy: Medication selection will be determined based on individual participant preferences, medical history, and contraindications. Options will include nicotine replacement therapy (nicotine patch, nicotine gum, nicotine lozenge), bupropion, or varenicline. Medications will be provided as mono-therapy or in combination.
- Total: Total of all reporting groups
Arm/Group | Tailored Intervention Group | Enhanced Standard of Care Group | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 29 | 55
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (11.5) | 58.5 (8.8) | 56.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 28 | 27 | 55
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 32 | 63
Nicotine dependence [Mean (Standard Deviation); unit: units on a scale] — Possible scores range from 0 to 11. Higher scores indicate greater levels of nicotine dependence.
  units on a scale | 5.6 (2.3) | 5.7 (2.1) | 5.7 (2.2)
Cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes/day] | 22.3 (10.3) | 27.2 (25.7) | 24.7 (19.4)
Prior quit attempts lasting at least 24 hours [Mean (Standard Deviation); unit: quit attempts] | 6.6 (8.1) | 9.4 (19.6) | 8.0 (15.0)
Readiness to quit smoking [Mean (Standard Deviation); unit: units on a scale] — Scores range from 1 to 10, with higher scores indicating greater readiness to quit smoking.
  units on a scale | 6.8 (1.1) | 6.5 (1.3) | 6.6 (1.2)
Age of smoking initiation [Mean (Standard Deviation); unit: years] | 16.7 (3.4) | 15.8 (2.8) | 16.2 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Satisfaction
Description: Participants' impressions of and satisfaction with the intervention will be assessed by interview at the end of treatment.
Time Frame: End of treatment (seven weeks after baseline)
Population: Participants who completed treatment satisfaction items on three-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Intervention Group | Enhanced Standard of Care Group
Number analyzed (Participants) | 23 | 14
Participants
  Found treatment very or extremely useful: number analyzed (Participants) | 23 | 13
  Found treatment very or extremely useful | 17 | 6
  Found medication to be very or extremely useful: number analyzed (Participants) | 21 | 13
  Found medication to be very or extremely useful | 16 | 7
  Found treatment to be very or extremely convenient: number analyzed (Participants) | 22 | 12
  Found treatment to be very or extremely convenient | 16 | 9
  Found treatment to be very or extremely difficult: number analyzed (Participants) | 20 | 11
  Found treatment to be very or extremely difficult | 5 | 5
  Liked that treatment was delivered by phone | 21 | 10

2. Secondary Outcome: Number of Participants Abstinent From Tobacco Use
Description: At the six-month follow-up contact, participants will be questioned regarding self-reported tobacco use over the past seven days (point prevalence abstinence).
Time Frame: Six-month follow-up
Population: 7-day point prevalence abstinence at 6 months. Those with missing data treated as smokers (penalized imputation).
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Intervention Group | Enhanced Standard of Care Group
Number analyzed (Participants) | 31 | 32
Participants | 9 | 9

3. Secondary Outcome: Alcohol Use
Description: Alcohol use during the previous seven days will be assessed among those receiving the risky alcohol use treatment module and those in the quitline referral condition who would have been eligible for the intervention if assigned to the tailored treatment group.
Time Frame: Six-month follow-up
Population: Participants in the tailored intervention group who received the alcohol intervention and those in the enhanced standard of care group who would have been eligible for the alcohol intervention if they had been assigned to the tailored intervention group.
Measure: Mean (Standard Deviation); unit: Drinks consumed per day
Arm/Group | Tailored Intervention Group | Enhanced Standard of Care Group
Number analyzed (Participants) | 2 | 4
Drinks consumed per day | 9.5 (0.7) | 2.8 (3.2)

4. Secondary Outcome: Depressive Symptoms
Description: Depressive symptoms as measured using the Patient Health Questionnaire 9 (PHQ-9). Possible scores range from 0 to 27, with higher scores indicating greater levels of depressive symptoms.
Time Frame: Six-month follow-up
Population: Participants in the tailored intervention group who receive the mood management module and those in the enhanced standard of care condition who would have been eligible for the mood management module if they had been assigned to the tailored intervention condition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored Intervention Group | Enhanced Standard of Care Group
Number analyzed (Participants) | 13 | 16
units on a scale | 7.0 (5.4) | 3.9 (2.7)

5. Secondary Outcome: Body Weight
Description: Self-reported body weight.
Time Frame: Six-month follow-up
Population: Assessed among participants in the tailored intervention group who received the weight management module and those in the enhanced standard of care condition who would have been eligible for the weight management module if they had been assigned to the tailored intervention condition.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Tailored Intervention Group | Enhanced Standard of Care Group
Number analyzed (Participants) | 6 | 9
Pounds | 214.0 (38.1) | 228.2 (45.5)

6. Secondary Outcome: Enrollment Rate
Description: The number of participants enrolled will be tracked as a measure of the feasibility of the intervention approached for the entire six-month recruitment period.
Time Frame: 6 months after study initiation
Population: Total number of participants randomized to each treatment condition.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Intervention Group | Enhanced Standard of Care Group
Number analyzed (Participants) | 31 | 32
Participants | 31 | 32

7. Secondary Outcome: Retention
Description: The number of participants who remain in the study throughout the seven-week treatment period will be computed as an indicator of the feasibility of the treatment approach.
Time Frame: End of treatment (seven weeks after baseline)
Population: Participants assigned to the tailored intervention condition who completed the intervention calls.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Intervention Group
Number analyzed (Participants) | 31
Participants | 16

8. Secondary Outcome: Treatment Attendance
Description: The number of treatment calls completed (out of six total) will be calculated for all participants in the Tailored Intervention group as an indicator of the feasibility of the treatment approach.
Time Frame: End of treatment (seven weeks after baseline)
Population: Attendance rate (number of counseling calls completed out of 6) among those assigned to the tailored intervention condition.
Measure: Mean (Full Range); unit: Calls
Arm/Group | Tailored Intervention Group
Number analyzed (Participants) | 31
Calls | 4.0 [0 to 6]

ADVERSE EVENTS:
Time Frame: Six months
Description: Data regarding adverse events were collected via self-report and information provided in patients' electronic medical record.
Arm/Group | Tailored Intervention Group | Enhanced Standard of Care Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 0/31 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No